CLINICAL TRIAL: NCT06128148
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of JYP0322 in Patients With Solid Tumors
Brief Title: Phase I Study of JYP0322 in ROS1 Fusion-Positive Solid Tumors
Acronym: JYP0322
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JYP0322M101
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-11

CONDITIONS: Protein Kinase Inhibitors; Other Protocol Specified Criteria; Lung Neoplasms; Brain Neoplasms
Keywords: ROS1 Fusions; ROS1 Gene Rearrangements; Primary brain tumors; ROS1
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms | interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 50 mg qd (Experimental): Participants with ROS1 fusion-positive locally advanced or metastatic solid tumors will receive JYP0322 at a dose of 50 mg qd. This arm evaluates the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of this dose level.
  Interventions: Drug: JYP0322 50 mg qd
- 100 mg qd (Experimental): Participants with ROS1 fusion-positive locally advanced or metastatic solid tumors will receive JYP0322 at a dose of 100 mg qd. This arm assesses safety, tolerability, and pharmacokinetics (PK) data for this dose level.
  Interventions: Drug: JYP0322 100 mg qd
- 200 mg qd (Experimental): Participants with ROS1 fusion-positive locally advanced or metastatic solid tumors will receive JYP0322 at a dose of 200 mg qd. This arm examines the safety, pharmacokinetics (PK), and preliminary efficacy of this dose level.
  Interventions: Drug: JYP0322 200 mg qd
- 100 mg bid (Experimental): Participants with ROS1 fusion-positive locally advanced or metastatic solid tumors will receive JYP0322 at a dose of 100 mg bid. The arm evaluates the safety, tolerability, and pharmacokinetics (PK) of this increased dosing frequency.
  Interventions: Drug: JYP0322 100 mg bid
- 150 mg bid (Experimental): Participants with ROS1 fusion-positive locally advanced or metastatic solid tumors will receive JYP0322 at a dose of 150 mg bid. This arm aims to determine the optimal dosing for safety, pharmacokinetics (PK), and efficacy.
  Interventions: Drug: JYP0322 150 mg bid
- 200 mg bid (Experimental): Participants with ROS1 fusion-positive locally advanced or metastatic solid tumors will receive JYP0322 at a dose of 200 mg bid. This arm focuses on evaluating safety, tolerability, and pharmacokinetics (PK) at this dose.
  Interventions: Drug: JYP0322 200 mg bid
- 150 mg tid (Experimental): Participants with ROS1 fusion-positive locally advanced or metastatic solid tumors will receive JYP0322 at a dose of 150 mg tid. This arm focuses on evaluating safety, tolerability, and pharmacokinetics (PK) at this dose.
  Interventions: Drug: JYP0322 150mg tid

INTERVENTIONS:
Drug: JYP0322 50 mg qd — JYP0322 is administered orally at a dose of 50 mg qd for a specified duration until unacceptable toxicity, disease progression, or study completion.
  Arms: 50 mg qd
Drug: JYP0322 100 mg qd — JYP0322 is administered orally at a dose of 100 mg qd for a specified duration until unacceptable toxicity, disease progression, or study completion.
  Arms: 100 mg qd
Drug: JYP0322 200 mg qd — JYP0322 is administered orally at a dose of 200 mg qd for a specified duration until unacceptable toxicity, disease progression, or study completion.
  Arms: 200 mg qd
Drug: JYP0322 100 mg bid — JYP0322 is administered orally at a dose of 100 mg bid for a specified duration until unacceptable toxicity, disease progression, or study completion.
  Arms: 100 mg bid
Drug: JYP0322 150 mg bid — JYP0322 is administered orally at a dose of 150 mg bid for a specified duration until unacceptable toxicity, disease progression, or study completion.
  Arms: 150 mg bid
Drug: JYP0322 200 mg bid — JYP0322 is administered orally at a dose of 200 mg bid for a specified duration until unacceptable toxicity, disease progression, or study completion.
  Arms: 200 mg bid
Drug: JYP0322 150mg tid — JYP0322 is administered orally at a dose of 150 mg tid for a specified duration until unacceptable toxicity, disease progression, or study completion.
  Arms: 150 mg tid

SUMMARY:
An open, non-randomized, multicenter, single-arm dose-escalation design, phase 1 trial to study the safety, tolerability, pharmacokinetics and efficacy of JYP0322 in patients with ROS1+ locally advanced/metastatic solid tumors .

DETAILED DESCRIPTION:
JYP0322 is an orally available inhibitor of ROS1 (coded by the gene ROS1). Molecular fusions are present in several different tumor types, including non-small cell lung cancer (NSCLC), glioma, etc. Patients with locally advanced or metastatic cancer with a detectable molecular fusion in targets of interest may be eligible for enrollment.

Phase 1 will assess safety and tolerability of JYP0322 via standard dose escalation scheme and determine the recommended Phase 2 dose. Safety and efficacy will be assessed in the dose expansion portion of the study.

ELIGIBILITY:
Key Inclusion Criteria

* Adult patients age 18 years or older.
* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumors that have a ROS1 molecular fusion.
* Measurable disease according to RECIST version 1.1
* Life expectancy of at least 3 months
* Other protocol specified criteria

Key Exclusion Criteria:

* Current participation in another therapeutic clinical trial.
* Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact on drug absorption.
* A history of severe allergies, or a history of severe allergy, hypersensitivity or other hypersensitivity to any active or inactive ingredient of the study drug.
* Known active infections (bacterial, viral including HIV positivity).
* Other protocol specified criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The frequency and severity of adverse events of JYP0322 | From the date of informed consent through 30 days after the last dose of study drug, approximately up to 36 months.
  Evaluate the safety and tolerability of JYP0322 treatment. This will be assessed by:
  Incidence, nature, and severity of adverse events (AEs) during treatment, the proportion of patients requiring dose adjustment or permanent drug discontinuation.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the first dose of study drug until disease progression, assessed by imaging every 8 weeks for the first 52 weeks, and every 12 weeks thereafter, up to 36 months.
  ORR is the proportion of subjects with CR or PR , based on RECIST v1.1 criteria.
Disease Control Rate (DCR) | From the first dose of study drug until disease progression, assessed by imaging every 8 weeks for the first 52 weeks, and every 12 weeks thereafter, up to 36 months.
  DCR is the proportion of subjects with CR or PR or SD, based on RECIST v1.1 criteria.
Duration of Response (DOR) | From the date of first response until disease progression or death, assessed by imaging every 8 weeks for the first 52 weeks, and every 12 weeks thereafter, up to 36 months.
  The time from the first documented objective response to the first occurrence of tumor progression or death from any cause.
Time to Response (TTR) | From the first dose of study drug to the date of first objective response, assessed by imaging every 8 weeks for the first 52 weeks, and every 12 weeks thereafter, up to 36 months.
  The time from treatment initiation to the first documented objective response.
Progression-Free Survival (PFS) | From the first dose of study drug until disease progression or death, assessed by imaging every 8 weeks for the first 52 weeks, and every 12 weeks thereafter, up to 36 months.
  The time from initiation of JYP0322 treatment to tumor progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No